CLINICAL TRIAL: NCT06420258
Title: A Study on the Effectiveness and Safety of Intratracheal Deep Intubation Compared to Traditional Tracheal Intubation in Endoscopic Submucosal Dissection for Early Esophageal Cancer in the Cervical Esophagus: A Randomized Controlled Trial.
Brief Title: Deeper Intubation Make Effects on Cervical Esophageal ESD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Wei Liang, Doctor, Fujian Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K2023-10-008
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Carcinoma in Situ of Cervical Part of Esophagus
Keywords: Deep tracheal intubation; Cervical esophageal cancer; ESD

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Each group allocation will be sealed in an opaque envelope with a code written on the outside. These sealed envelopes will be handed over to the researchers. When a study participant meets the inclusion and exclusion criteria upon entry into the study, they will be assigned a number. Subsequently, the corresponding envelope with the assigned number will be opened, and the intervention will be carried out according to the group allocation specified in the envelope. The treatment plan for each research participant will be determined by the generated random sequence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deeper endotracheal intubation (Experimental): After general anesthesia, endotracheal intubation was conducted using an ultrafine endoscope (GIF-XP260NS, Olympus Corp., Japan), which allows observation of the exact position and avoids blindness caused by laryngoscopy. To prevent balloon compression of the CE after inflating, the endotracheal intubation tube was inserted above the tracheal carina, roughly the upper thoracic esophagus
  Interventions: Procedure: Deeper endotracheal intubation
- Conventional endotracheal intubation (No Intervention)

INTERVENTIONS:
Procedure: Deeper endotracheal intubation — After general anesthesia, endotracheal intubation was conducted using an ultrafine endoscope (GIF-XP260NS, Olympus Corp., Japan), which allows observation of the exact position and avoids blindness caused by laryngoscopy. To prevent balloon compression of the CE after inflating, the endotracheal intubation tube was inserted above the tracheal carina, roughly the upper thoracic esophagus.
  Arms: Deeper endotracheal intubation

SUMMARY:
To compare the efficacy and safety of intratracheal deep intubation with traditional intubation in endoscopic submucosal dissection for early esophageal cancer in the cervical esophagus, and to follow up and assess their short-term clinical outcomes.

DETAILED DESCRIPTION:
Forty patients with early esophageal cancer in the cervical esophagus scheduled for endoscopic submucosal dissection will be included. They will be randomly divided into two groups using sealed envelopes: approximately 20 patients in the intratracheal deep intubation group and 20 patients in the traditional intubation group. By comparing the operation time, perioperative complications, postoperative short-term complications, and other outcomes, we aim to elucidate the effectiveness and safety of deep intubation in endoscopic submucosal dissection for early esophageal cancer in the cervical esophagus.

ELIGIBILITY:
Inclusion Criteria:

1. The lesions mainly involve superficial esophageal squamous cell carcinoma or high-grade intraepithelial neoplasia (HGIN) in the cervical esophagus;
2. There is no evidence of regional lymph node or distant metastasis on endoscopic ultrasound (EUS) or CT/MRI imaging;
3. Participants have a thorough understanding of this study and voluntarily sign the informed consent form.

Exclusion Criteria:

* 1. Patients who have received radiotherapy or chemotherapy before endoscopic submucosal dissection surgery; 2. Patients with severe comorbidities who are not suitable for endoscopic submucosal dissection surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the rate of complete resection and postoperative stricture | Seven days and three months after ESD procedure

SECONDARY OUTCOMES:
ESD procedural time and other procedure-related complications | During procedures and just after ESD procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Liang, MD, Study Director — Fujian Provintial Hospital
Locations (1):
- Fujian Provintial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu Y, Wu Y, Deng W, Guo X, Gao P, Yang S, Chen Y, Zhou P, Liang W. More efficient endoscopic submucosal dissection with deep endotracheal intubation for superficial cervical esophageal carcinoma: a dual-center, prospective, randomized controlled study. Gastrointest Endosc. 2025 Mar;101(3):655-658. doi: 10.1016/j.gie.2024.09.018. Epub 2024 Sep 13. PMID 39278284